CLINICAL TRIAL: NCT01425892
Title: The Pathogenesis and Natural History of Sjogren's Disease
Status: Recruiting | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110172; 11-D-0172
Record Dates: First submitted 2011-08-27; First posted 2011-08-30 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01-20

CONDITIONS: Sjogren's Syndrome; Salivary Gland; Pathogenesis
Keywords: Sjogren's Syndrome; Salivary Gland; Pathogenesis; Natural History; Sj(SqrRoot)(Delta)gren s syndrome; Sjogrens Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- incomplete sjogren's: patients who meet criteria as incomplete sjogren's
- primary sjogren's: patients who meet criteria for classification for primary sjogren's
- secondary sjogren's: patients who meet classification criteria for secondary sjogren's

SUMMARY:
Background:

-Sjogren s Disease (formerly: Sjogrens Syndrome, Sj(SqrRoot)(Delta)gren s syndrome) is a disease that affects about 1-4 million Americans. It is more common in women. It mainly affects the glands that produce saliva and tears, leading to dry eyes and dry mouth. The cause of Sjogren s Disease is unknown, but inflammation plays an important role. The purpose of this study is to learn more about Sjogren s Disease.

Objectives:

-To better understand how Sjogren s Disease begins and how it affects patients so that we can develop better ways to treat them.

Eligibility:

* Participants must be 16 years of age or older.
* They must have a diagnosis of Sjogren s Disease or have at least two symptoms of Sjogren s Disease.

Design:

* People taking part in the study will come to the NIH Clinical Center for at least three visits.
* During these visits, participants will have a medical history and physical exam. They will have oral and dental assessments, and saliva collection. Lab tests (blood and urine) and dry eye exams will be done. Participants will answer questionnaires and have salivary scintigraphy (adults only unless required for diagnosis).
* Other optional tests may also be done. Participants may have to come in for additional visits if they have these optional tests or if their disease changes.
* The only treatment provided as part of this study is for medical emergencies or complications that occur while you are at NIH for evaluation.

DETAILED DESCRIPTION:
Background

Sjogren's Disease (SjD; formely Sjogren's Syndrome) is an autoimmune disease characterized by chronic inflammation involving the exocrine glands. Salivary and lacrimal glands are predominantly affected leading to dry mouth and dry eyes but other exocrine organs are also frequently involved. It is one of the most common rheumatic autoimmune diseases, which effects between 1-4 million Americans, predominantly women with a female to male ratio of 9:1. Sjogren s Disease may occur alone (primary SjD), or may coexist with other systemic connective tissue disorders (i.e., secondary SjD). In many cases systemic manifestations, such as fatigue, arthritis, vasculitis, lung disease, peripheral or central neuropathy and autonomic nervous system dysfunction accompany glandular involvement. Patients with systemic manifestations are at higher risk of lymphoma, the incidence of which is increased in SjD. The treatment of sicca symptoms is mainly symptomatic, whereas management of extraglandular manifestations is similar to other autoimmune diseases.

The cause and pathogenesis of Sjogren's Disease is still largely unknown. In a genetically predisposed individual various environmental factors, such as viral infections, may lead to epithelial cell activation and a protracted inflammatory response with features of autoimmunity. Autoreactive lymphocytes and autoantibodies are considered important in this process although the pathogenic role of any particular autoantibody is still undefined. Although inflammation may contribute to the exocrinopathy of SjD, the relationship between inflammation and exocrine dysfunction is poorly understood. Moreover, the model does not explain many of the extraglandular manifestations of SjD patients, such as fatigue. Further studies are needed to better understand the pathogenesis of SjD.

Objectives

The primary objective of this study is to enable the collection of longitudinal clinical and laboratory data and biologic specimens to identify pathogenetic mechanisms of SjD by careful clinical phenotyping of SjD patients and Sjogren's-like conditions over time and collection of biologic samples for concurrent and future laboratory studies related to the pathogenesis of Sjogren's Disease. Another objective of the study is to identify biomarker candidates associated with the diagnosis, severity, prognosis, or organ involvement in SjD. The protocol will enable the study of the genetic basis and the mechanistic aspects of immunologic and non-immunologic abnormalities of SjD and their associations with various clinical phenotypes.

Eligibility Criteria

The study will enroll 300 subjects with Sjogren s Disease or Sjogren's-like conditions. Subjects aged 16-years or older fulfilling European American Consensus Criteria for Primary or Secondary Sjogren s Disease are eligible for the study. Selected subjects with incomplete Sjogren's Disease or who are excluded from the European American criteria may also be eligible. Screening will be done on the Characterization of Diseases with Salivary Gland Involvement protocol (15-D-0051) prospectively or on the previous screening protocol (84-D-0056).

Description of the Study

This is a longitudinal observational study. All subjects will have core evaluations (approximately biannually) during a 10-year period. Additional evaluations may be required if there is a significant change in the clinical condition of subjects likely related to SjD or sicca syndrome or to provide additional research samples or clinical data for the pathogenesis studies. Clinical data will be collected through questionnaires, personal interviews, physical examination, laboratory testing and imaging studies. The core evaluation will include a complete medical history and physical examination and a complete oral and dry eye evaluation. Blood, saliva and biopsy samples will be stored and used for laboratory research studies aimed at the pathogenesis of Sjogren s Disease. Samples labeled with a code without any personal identifiers may be shared with researchers in and outside the NIH. DNA will be collected for genetic studies related to Sjogren's' syndrome and related conditions.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Ability to sign informed consent form
  2. Fulfilling one the definitions below:

     1. Sjogren s defined by European-American (EA) classification criteria for primary or secondary Sjogren s Disease (SjD group)
     2. Excluded from the EA criteria because of a comorbid condition but otherwise fulfilling the European-American classification criteria (EA excluded SjD group)
     3. Incomplete SjD

     i. at least 2 of the EA criteria with a common manifestation of SjD not included in these criteria (e.g., fatigue, vasculitis, arthritis, etc) or

     ii. 2 or more common manifestations of SjD which are not included in the EA criteria (e.g.,: fatigue, vasculitis, arthritis, autonomic dysfunction, etc ) and are not explained by other conditions

     EXCLUSION CRITERIA:

  <!-- -->

  1. Age <16 years
  2. inability or unwillingness to comply with follow up requirements
  3. Any medical or psychological/psychiatric condition or treatment that, in the opinion of the Principal Investigator, would exclude the subjects from the research studies (e.g., alternative explanation for subjects signs and symptoms)
  4. NIH employees who report directly to the principal investigator or who are a co-worker or relative of the principal investigator.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population consists of patients who have completed our Sjogren's screening protocol (15-D-0051) and are deemed eligible to enroll in this pathogenesis protocol.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-01-18 (Actual)

PRIMARY OUTCOMES:
Clinical phenotyping of SjD patients and controls over time Collection of samples for concurrent and future laboratory studies related to the pathogenesis Identification of biomarker candidates in SjD | patients are followed up to 10 years
  following the natural history of Sjogren's disease progression.

SECONDARY OUTCOMES:
1. To establish a teaching cohort of patients with SjD or SjD-like conditions treated with conventional treatments 2. To identify patients for other protocols related to Sjogren's Disease | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Zohreh Khavandgar, D.D.S., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This is a natural history study that began enrolling in 2011. De-identified data will be made public consistent with the policies of the NIH.

REFERENCES:
- [Derived] Burbelo PD, Ferre EMN, Chaturvedi A, Chiorini JA, Alevizos I, Lionakis MS, Warner BM. Profiling Autoantibodies against Salivary Proteins in Sicca Conditions. J Dent Res. 2019 Jul;98(7):772-778. doi: 10.1177/0022034519850564. Epub 2019 May 16. PMID 31095438
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-D-0172.html